CLINICAL TRIAL: NCT00771394
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study of Solifenacin Succinate as Add-on Therapy for Overactive Bladder (OAB) Symptoms in Men Treated for Benign Prostatic Hyperplasia (BPH) With Tamsulosin Hydrochloride
Brief Title: Solifenacin as Add-on Therapy for Overactive Bladder Symptoms in Men Treated for Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 905-JC-001
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Benign Prostatic Hyperplasia; Benign Prostatic Hypertrophy; Overactive Bladder
Keywords: Vesicare; Solifenacin succinate; Tamsulosin; Overactive Bladder; BPH
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder, Overactive | interventions — Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. Tamsulosin alone (Placebo Comparator)
  Interventions: Drug: Tamsulosin hydrochloride
- 2. Tamsulosin + solifenacin (low dose) (Experimental)
  Interventions: Drug: Tamsulosin hydrochloride; Drug: Solifenacin succinate
- 3. Tamsulosin + solifenacin (high dose) (Active Comparator)
  Interventions: Drug: Tamsulosin hydrochloride; Drug: Solifenacin succinate

INTERVENTIONS:
Drug: Tamsulosin hydrochloride — oral
  Other Names: Harnal; YM617
Drug: Solifenacin succinate — oral
  Other Names: Vesicare; YM905
  Arms: 2. Tamsulosin + solifenacin (low dose); 3. Tamsulosin + solifenacin (high dose)

SUMMARY:
To evaluate the efficacy and safety of solifenacin succinate as add-on therapy for overactive bladder (OAB) symptoms in men who have been treated for benign prostatic hyperplasia (BPH) with tamsulosin hydrochloride for at least 6 weeks

DETAILED DESCRIPTION:
Study drugs are administered for 14 weeks in total, including a 2-week run-in period (single blind) and a 12-week treatment period (double blind). After written informed consent, study drugs for the run-in period are orally administered once daily after breakfast for two weeks to subjects who fulfill the inclusion and exclusion criteria. Then, subjects are randomized and orally treated with study drugs for the treatment period once daily after breakfast for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign prostatic hypertrophy who have been treated with tamsulosin for at least 6 weeks
* Patients with urgency episodes and frequent micturitions
* Written informed consent has been obtained
* Uroflowmetry-Q max ≥ 5 mL/sec, and Post Void Residual Volume < 50 mL

Exclusion Criteria:

* Patients with suspected symptoms of OAB whose onset is only transient (drug-induced, psychogenic, etc.)
* Patients with obvious stress urinary incontinence
* Patients with complications or who have a past history of a bladder tumor
* Patients with urethral stricture or bladder neck stenosis
* Patients with a history of surgery causing damage to the pelvic plexus
* Patients with history of hypersensitivity to α receptor blockers, a/b receptor blockers, or anticholinergic drugs
* Patients with orthostatic hypotension, ulcerative colitis, hyperthyroidism, dementia or cognitive dysfunction, Parkinson's disease, or cerebrovascular disorder

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean number of urgency episodes per 24 hours | at 4, 8, 12 week

SECONDARY OUTCOMES:
Mean number of micturitions per 24 hrs | at 4, 8, 12 week
Mean number of incontinence episodes per 24 hours | at 4, 8, 12 week
Mean number of micturitions per night | at 4, 8, 12 week
Adverse Events, Laboratory Tests | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku